CLINICAL TRIAL: NCT02490995
Title: Inform and Reduce Pre-surgical Anxiety of the Child and His Parents: Interest of an Explanatory Movie About the Pathway of the Child in Pediatric Surgery.
Brief Title: Inform and Reduce Pre-surgical Anxiety of the Child and His Parents: Interest of an Explanatory Movie.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9392; 2014-A00416-41 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Anxiety Linked to the Surgery and / or Anesthesia
Keywords: children
MeSH Terms: interventions — Motion Pictures

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (No Intervention): Information given by the anaesthetist during the consultation
- Group B (Experimental): Movie + Information given by the anaesthetist during the consultation
  Interventions: Other: Movie

INTERVENTIONS:
Other: Movie — Besides the anesthesist explanations the children will have a movie explanation.
  Arms: Group B

SUMMARY:
The purpose of the study is to measure the interest of a movie explaining the path of the children in surgery, in order to reduce the anxiety of the children and his parents.

This study is interventional, method randomized, controled, open-label, comparing two parallel arms: anesthesist explanations versus anesthesist explanations + a movie explanation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who need a surgery
* Patient that general condition fit with American Society of Anesthesiologists (ASA) I to III classification.
* Old patient under age 12
* Patient whose parents agreed to participate

Exclusion Criteria:

* Patient with psychomotor limitations
* Patient that had already been hospitalised for a surgery

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The Yale Preoperative Anxiety Scale (m-YPAS) | the 1 surgery day at the time of the separation parents-children
  Pre-surgical anxiety score of the children when separate from his parents, measured with the Yale Preoperative Anxiety Scale (m-YPAS)

SECONDARY OUTCOMES:
Induction Compliance Checklist (ICC) | intraoperative
  Score of "compliance" in the anesthetic induction measured by the ICC scale (hetero-assessment)
The agitation in recovery room | First 15 minutes of the arrival in recovery room
  The agitation in recovery room measured by the scale of agitation in the awakening of a pediatric anesthesia (EPAD) (hetero-assessment)
psychometric validation of the SAS (self anxiety scale) | up to postoperative day 30
  validation of the self report anxiety scale

CONTACTS AND LOCATIONS:
Overall Officials: Sophie SB Bringuier, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier university hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified data used in the published manuscript will be shared in accordance with the applicable informed consent under which the data was collected
  Supporting Information:
  Time Frame:
  12 months after the main publication
  Access Criteria:
  Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and IRB review. Dataset will be shared after careful examination by the study board of investigators.
  Identified data used in the published manuscript will be shared in accordance with the applicable informed consent under which the data was collected
  Supporting Information:
Supporting Information: CSR
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and IRB review. Dataset will be shared after careful examination by the study board of investigators.